CLINICAL TRIAL: NCT05140239
Title: Effects of Abrocitinib Treatment of Moderate to Severe Atopic Dermatitis on Skin Barrier Function
Brief Title: Effects of Abrocitinib Treatment on Skin Barrier Function
Acronym: AbroSkib
Status: Active, not recruiting | Type: Observational
Sponsor: Prof. Dr. Stephan Weidinger (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Stephan Weidinger, Vice Head, Department of Dermatology and Allergy, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Other Study IDs: ABRO_WEI_2021
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Atopic Dermatitis
Keywords: Skin Barrier; Atopic Dermatitis; Dermatology; Skin Physiology
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin swabs, tape strips.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AbroSkib Cohort: Adult patients with moderate to severe atopic dermatitis who are eligible for and will receive systemic therapy with abrocitinib by their treating dermatologist as part of standard healthcare (n=20). The choice of therapy is strictly done by the treating dermatologist only, and the reasons for the choice will be captured by a structured documentation.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Non Interventional

SUMMARY:
Effects of abrocitinib treatment of atopic dermatitis on skin barrier function.

DETAILED DESCRIPTION:
Open-label, non-randomized, single-arm, 12-weeks observational clinical and translational study

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related pro-cedures, including screening evaluations
2. Age ≥ 18 years at time of study entry.
3. Diagnosis of chronic atopic dermatitis for at least 1 year prior to enrollment based on American Academy Criteria
4. Eczema Area and Severity Index (EASI) score ≥12 at baseline visit (Week 0)
5. Investigator Global Assessment (IGA) ≥3 at baseline visit (Week 0)
6. Subject is willing and able to comply with the protocol for the duration of the study
7. Subject receives abrocitinib by the treating dermatologist within routine care

Exclusion Criteria:

1. 1. Subject is unable to provide written informed consent or comply with the protocol
2. Concurrent enrolment in another clinical trial where the subject is receiving an IMP or participation in another clinical trial with investigational product during the last 30 days before inclusion or 7 half-lives of previously used trial medication, whichever is longer.
3. Active dermatologic conditions that may confound the diagnosis of AD or would interfere with as-sessment of treatment, such as scabies, cutaneous lymphoma, or psoriasis.
4. Known active allergic or irritant contact dermatitis that is likely to interfere with the assessment of severity of AD.
5. Having used systemic immunosuppressive/immunomodulating therapy (e.g. systemic corticoster-oids methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, JAK inhibitors) or tanning beds or phototherapy during any week within the 4 weeks or receipt of any marketed biologic ther-apy (e.g., dupilumab, tralokinumab) within 3 months or 5 half-lives, whichever is longer, prior to baseline
6. Treatment of selected marker skin areas (non-lesional skin at volar forearm and extensor forearm, lesional skin) with topical corticosteroid or topical calcineurin inhibitor 1 week prior to baseline visit and throughout the study.
7. Treatment of skin areas of examination with emollients 24 hours prior to baseline visit and throughout the study.
8. Involvement in the planning and/or conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (n=20) with moderate to severe atopic dermatitis who are eligible for and will receive systemic therapy with abrocitinib by their treating dermatologist as part of standard healthcare. The choice of therapy is strictly done by the treating dermatologist only, and the reasons for the choice will be captured by a structured documentation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in transepidermal water loss (TEWL) at one non-lesional and one lesional marker skin area at week 2 and week 12 compared to baseline/week 0 (day 0). | 12 Weeks
  To determine the mean change of TEWL in g/m2/h at one non-lesional and one lesional marker skin site at week 2 and week 12 compared to baseline

SECONDARY OUTCOMES:
Number of epidermal barrier-related genes/pathways differentially expressed in a marker lesional skin site at week 2 and week 12 compared to baseline | 12 Weeks
  To compare the expression of epidermal barrier-related genes at the transcriptome level at a marker lesional skin site at week 2 and week 12 to baseline and to non-lesional skin
Epidermal thickness and epidermal differentiation markers in a marker lesional skin site at week 2 and week 12 compared to baseline | 12 Weeks
  To compare epidermal thickness (in µm) and the percentage of marker-positive cells (KRT 16, Ki67, FLG) in a marker skin site with reference to the number of cells in the basal layer at week 2 and 12 to baseline and to non-lesional skin
Stratum corneum biomarker (cytokine) levels (pg/μg protein) in marker skin sites at week 2 and week 12 compared to baseline | 12 Weeks
  To compare stratum corneum biomarker (cytokine) levels (pg/μg protein) in a marker lesional skin site at week 2 and week 12 compared to baseline and to non-lesional skin
Composition of Bacterial Taxa of one lesional and non-lesional marker skin area at week 2 and week 12 compared to baseline | 12 Weeks
  To identify changes in community composition and diversity at one lesional and one non-lesional marker skin site at week 2 and week 12 as compared to baseline using Next Generation Sequencing techniques

OTHER OUTCOMES:
Transcriptional profile of the keratinocytes in one lesional marker skin area at week 2 and 12 compared to baseline | 12 Weeks
  To compare the transcriptional profile of keratinocytes at one lesional marker skin area at week 2 and 12 compared to baseline and to non-lesional skin using single cell sequencing techniques

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, MD, Principal Investigator — UKSH Kiel, University of Kiel
Locations (1):
- UKSH, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langan SM, Irvine AD, Weidinger S. Atopic dermatitis. Lancet. 2020 Aug 1;396(10247):345-360. doi: 10.1016/S0140-6736(20)31286-1. PMID 32738956
- [Background] Moitinho-Silva L, Boraczynski N, Emmert H, Baurecht H, Szymczak S, Schulz H, Haller D, Linseisen J, Gieger C, Peters A, Tittmann L, Lieb W, Bang C, Franke A, Rodriguez E, Weidinger S. Host traits, lifestyle and environment are associated with human skin bacteria. Br J Dermatol. 2021 Sep;185(3):573-584. doi: 10.1111/bjd.20072. Epub 2021 May 18. PMID 33733457
- [Background] Tsoi LC, Rodriguez E, Stolzl D, Wehkamp U, Sun J, Gerdes S, Sarkar MK, Hubenthal M, Zeng C, Uppala R, Xing X, Thielking F, Billi AC, Swindell WR, Shefler A, Chen J, Patrick MT, Harms PW, Kahlenberg JM, Perez White BE, Maverakis E, Gudjonsson JE, Weidinger S. Progression of acute-to-chronic atopic dermatitis is associated with quantitative rather than qualitative changes in cytokine responses. J Allergy Clin Immunol. 2020 May;145(5):1406-1415. doi: 10.1016/j.jaci.2019.11.047. Epub 2019 Dec 28. PMID 31891686
- [Background] Tsoi LC, Rodriguez E, Degenhardt F, Baurecht H, Wehkamp U, Volks N, Szymczak S, Swindell WR, Sarkar MK, Raja K, Shao S, Patrick M, Gao Y, Uppala R, Perez White BE, Getsios S, Harms PW, Maverakis E, Elder JT, Franke A, Gudjonsson JE, Weidinger S. Atopic Dermatitis Is an IL-13-Dominant Disease with Greater Molecular Heterogeneity Compared to Psoriasis. J Invest Dermatol. 2019 Jul;139(7):1480-1489. doi: 10.1016/j.jid.2018.12.018. Epub 2019 Jan 11. PMID 30641038
- [Background] Mobus L, Rodriguez E, Harder I, Stolzl D, Boraczynski N, Gerdes S, Kleinheinz A, Abraham S, Heratizadeh A, Handrick C, Haufe E, Werfel T, Schmitt J, Weidinger S; TREATgermany study group. Atopic dermatitis displays stable and dynamic skin transcriptome signatures. J Allergy Clin Immunol. 2021 Jan;147(1):213-223. doi: 10.1016/j.jaci.2020.06.012. Epub 2020 Jun 29. PMID 32615169
- [Background] Weidinger S, Beck LA, Bieber T, Kabashima K, Irvine AD. Atopic dermatitis. Nat Rev Dis Primers. 2018 Jun 21;4(1):1. doi: 10.1038/s41572-018-0001-z. PMID 29930242
- [Background] Thaci D, Simpson EL, Beck LA, Bieber T, Blauvelt A, Papp K, Soong W, Worm M, Szepietowski JC, Sofen H, Kawashima M, Wu R, Weinstein SP, Graham NM, Pirozzi G, Teper A, Sutherland ER, Mastey V, Stahl N, Yancopoulos GD, Ardeleanu M. Efficacy and safety of dupilumab in adults with moderate-to-severe atopic dermatitis inadequately controlled by topical treatments: a randomised, placebo-controlled, dose-ranging phase 2b trial. Lancet. 2016 Jan 2;387(10013):40-52. doi: 10.1016/S0140-6736(15)00388-8. Epub 2015 Oct 8. PMID 26454361
- [Background] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Background] Blauvelt A, de Bruin-Weller M, Gooderham M, Cather JC, Weisman J, Pariser D, Simpson EL, Papp KA, Hong HC, Rubel D, Foley P, Prens E, Griffiths CEM, Etoh T, Pinto PH, Pujol RM, Szepietowski JC, Ettler K, Kemeny L, Zhu X, Akinlade B, Hultsch T, Mastey V, Gadkari A, Eckert L, Amin N, Graham NMH, Pirozzi G, Stahl N, Yancopoulos GD, Shumel B. Long-term management of moderate-to-severe atopic dermatitis with dupilumab and concomitant topical corticosteroids (LIBERTY AD CHRONOS): a 1-year, randomised, double-blinded, placebo-controlled, phase 3 trial. Lancet. 2017 Jun 10;389(10086):2287-2303. doi: 10.1016/S0140-6736(17)31191-1. Epub 2017 May 4. PMID 28478972
- [Background] Abraham S, Haufe E, Harder I, Heratizadeh A, Kleinheinz A, Wollenberg A, Weisshaar E, Augustin M, Wiemers F, Zink A, Biedermann T, von Kiedrowski R, Hilgers M, Worm M, Pawlak M, Sticherling M, Fell I, Handrick C, Schakel K, Staubach P, Asmussen A, Schwarz B, Bell M, Neubert K, Effendy I, Bieber T, Homey B, Gerlach B, Tchitcherina E, Stahl M, Schwichtenberg U, Rossbacher J, Buck P, Mempel M, Beissert S, Werfel T, Weidinger S, Schmitt J; TREATgermany study group. Implementation of dupilumab in routine care of atopic eczema: results from the German national registry TREATgermany. Br J Dermatol. 2020 Aug;183(2):382-384. doi: 10.1111/bjd.18958. Epub 2020 Apr 13. No abstract available. PMID 32068242
- [Background] Gadina M, Le MT, Schwartz DM, Silvennoinen O, Nakayamada S, Yamaoka K, O'Shea JJ. Janus kinases to jakinibs: from basic insights to clinical practice. Rheumatology (Oxford). 2019 Feb 1;58(Suppl 1):i4-i16. doi: 10.1093/rheumatology/key432. PMID 30806710
- [Background] Simpson EL, Sinclair R, Forman S, Wollenberg A, Aschoff R, Cork M, Bieber T, Thyssen JP, Yosipovitch G, Flohr C, Magnolo N, Maari C, Feeney C, Biswas P, Tatulych S, Valdez H, Rojo R. Efficacy and safety of abrocitinib in adults and adolescents with moderate-to-severe atopic dermatitis (JADE MONO-1): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet. 2020 Jul 25;396(10246):255-266. doi: 10.1016/S0140-6736(20)30732-7. PMID 32711801
- [Background] Clarysse K, Pfaff CM, Marquardt Y, Huth L, Kortekaas Krohn I, Kluwig D, Luscher B, Gutermuth J, Baron J. JAK1/3 inhibition preserves epidermal morphology in full-thickness 3D skin models of atopic dermatitis and psoriasis. J Eur Acad Dermatol Venereol. 2019 Feb;33(2):367-375. doi: 10.1111/jdv.15301. Epub 2019 Jan 1. PMID 30357932
- [Background] Bieber T. Atopic dermatitis. Ann Dermatol. 2010 May;22(2):125-37. doi: 10.5021/ad.2010.22.2.125. Epub 2010 May 17. PMID 20548901
- [Background] Weidinger S, Novak N. Atopic dermatitis. Lancet. 2016 Mar 12;387(10023):1109-1122. doi: 10.1016/S0140-6736(15)00149-X. Epub 2015 Sep 13. PMID 26377142
- [Background] Silverberg JI, Hanifin JM. Adult eczema prevalence and associations with asthma and other health and demographic factors: a US population-based study. J Allergy Clin Immunol. 2013 Nov;132(5):1132-8. doi: 10.1016/j.jaci.2013.08.031. Epub 2013 Oct 4. PMID 24094544
- [Background] Kiebert G, Sorensen SV, Revicki D, Fagan SC, Doyle JJ, Cohen J, Fivenson D. Atopic dermatitis is associated with a decrement in health-related quality of life. Int J Dermatol. 2002 Mar;41(3):151-8. doi: 10.1046/j.1365-4362.2002.01436.x. PMID 12010340
- [Background] Emmert H, Baurecht H, Thielking F, Stolzl D, Rodriguez E, Harder I, Proksch E, Weidinger S. Stratum corneum lipidomics analysis reveals altered ceramide profile in atopic dermatitis patients across body sites with correlated changes in skin microbiome. Exp Dermatol. 2021 Oct;30(10):1398-1408. doi: 10.1111/exd.14185. Epub 2020 Sep 17. PMID 32885529
- [Background] Baurecht H, Ruhlemann MC, Rodriguez E, Thielking F, Harder I, Erkens AS, Stolzl D, Ellinghaus E, Hotze M, Lieb W, Wang S, Heinsen-Groth FA, Franke A, Weidinger S. Epidermal lipid composition, barrier integrity, and eczematous inflammation are associated with skin microbiome configuration. J Allergy Clin Immunol. 2018 May;141(5):1668-1676.e16. doi: 10.1016/j.jaci.2018.01.019. Epub 2018 Feb 5. PMID 29421277
- [Background] Suarez-Farinas M, Ungar B, Correa da Rosa J, Ewald DA, Rozenblit M, Gonzalez J, Xu H, Zheng X, Peng X, Estrada YD, Dillon SR, Krueger JG, Guttman-Yassky E. RNA sequencing atopic dermatitis transcriptome profiling provides insights into novel disease mechanisms with potential therapeutic implications. J Allergy Clin Immunol. 2015 May;135(5):1218-27. doi: 10.1016/j.jaci.2015.03.003. Epub 2015 Mar 31. PMID 25840722
- [Background] Welsch K, Holstein J, Laurence A, Ghoreschi K. Targeting JAK/STAT signalling in inflammatory skin diseases with small molecule inhibitors. Eur J Immunol. 2017 Jul;47(7):1096-1107. doi: 10.1002/eji.201646680. Epub 2017 Jun 21. PMID 28555727
- [Background] Guttman-Yassky E, Bissonnette R, Ungar B, Suarez-Farinas M, Ardeleanu M, Esaki H, Suprun M, Estrada Y, Xu H, Peng X, Silverberg JI, Menter A, Krueger JG, Zhang R, Chaudhry U, Swanson B, Graham NMH, Pirozzi G, Yancopoulos GD, D Hamilton JD. Dupilumab progressively improves systemic and cutaneous abnormalities in patients with atopic dermatitis. J Allergy Clin Immunol. 2019 Jan;143(1):155-172. doi: 10.1016/j.jaci.2018.08.022. Epub 2018 Sep 5. PMID 30194992
- [Background] Retzler J, Smith A, Reaney M, Rout R, Hudson R. Process utilities for topical treatment in atopic dermatitis. Qual Life Res. 2019 Sep;28(9):2373-2381. doi: 10.1007/s11136-019-02174-0. Epub 2019 Apr 3. PMID 30945132
- [Background] Danby SG, Chalmers J, Brown K, Williams HC, Cork MJ. A functional mechanistic study of the effect of emollients on the structure and function of the skin barrier. Br J Dermatol. 2016 Nov;175(5):1011-1019. doi: 10.1111/bjd.14684. Epub 2016 Aug 23. PMID 27097823
- See also: German Guidelines on Atopic Dermatitis — https://register.awmf.org/de/leitlinien/detail/013-027